CLINICAL TRIAL: NCT05625776
Title: Effects of Acute Pain on Cognitive Performance in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susanne M Morton, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1786370-1.2; R01AG071585 (NIH)
Record Dates: First submitted 2022-11-13; First posted 2022-11-23 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Pain, Acute; Cognition
Keywords: acute pain; cognition; pain; cognitive ability; young adults
MeSH Terms: conditions — Acute Pain; Pain | interventions — Capsaicin; Hot Temperature

STUDY DESIGN:
Masking Description: Application of pain or attentional control or no stimulus cannot be masked from participants, nor from outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Stimulus (Experimental): Capsaicin combined with heat applied to intact skin
  Interventions: Procedure: pain delivery with capsaicin and heat
- Distractor Somatosensory Stimulus (Active Comparator): Sensory transcutaneous electrical nerve stimulation (TENS) applied to intact skin
  Interventions: Procedure: distractor delivery with sensory TENS
- No Stimulus (No Intervention): Nothing applied to skin

INTERVENTIONS:
Procedure: pain delivery with capsaicin and heat — Experimental pain paradigm delivered (capsaicin cream combined with heat) that is short-term and painful but not harmful
  Arms: Pain Stimulus
Procedure: distractor delivery with sensory TENS — Distractor stimulus delivered (sensory TENS electrical stimulation) that is short-term and attention-demanding but not painful
  Arms: Distractor Somatosensory Stimulus

SUMMARY:
The effects of pain on cognitive performance have not been thoroughly investigated. Broadly, the purpose of this research is to investigate the effects of acute pain on performance of a variety of cognitive performance measures. The investigators hypothesize that acute pain impairs cognitive performance, particularly cognitive measures of working memory, attention, and processing speed.

ELIGIBILITY:
Abbreviations: HR= heart rate, bpm= beats per minute; BP= blood pressure; ADD= attention deficit disorder; ADHD= attention deficit hyperactivity disorder; MoCA= Montreal Cognitive Assessment; GAD-7= Generalized Anxiety Disorder 7 Scale; PHQ-2, PHQ-9= Patient Health Questionnaire-2 and -9.

Inclusion Criteria:

1. 18-35 years old
2. Self-identifying as generally medically healthy
3. Able to read, write and speak English
4. Able to provide informed consent
5. Willing to undergo the experimental pain or non-painful electrical stimulation, if selected

Exclusion Criteria:

1. Resting HR < 50 or > 100 bpm
2. Resting BP < 90/60 or > 140/95 mmHg
3. Any history or current mental health condition, learning/developmental disability or cognitive impairment, including ADD/ADHD, severe anxiety, severe depression, autism spectrum disorder, insomnia, mild cognitive impairment, etc.
4. Score on the MoCA <23
5. Score on the GAD-7 ≥ 10
6. Score on the PHQ-2 ≥ 2 and score on the PHQ-9 ≥ 10
7. Any current (within last 3 month) or chronic medical conditions, including any musculoskeletal, cardiovascular, endocrine, pulmonary, metabolic, psychiatric or neurological diagnosis
8. Any implanted electronic medical devices (i.e., cardiac pacemakers, cardiac defibrillators, spinal cord neurostimulators)
9. Any impaired sensation or weakness in either lower extremity or in the area targeted for the stimulus
10. History of serious concussion or head injury, defined as a loss of consciousness for > 5 minutes and/or requiring medical treatment, or > 2 concussions over the lifespan
11. Any history of acute or chronic problems with balance, any dizziness, or > 1 fall in the last 12 months
12. Taking 4 or more medications
13. Currently or regularly using any analgesic medications, over-the-counter remedies, or any other treatment for the purposes of pain relief (i.e., baby aspirin for heart health permitted, etc.)
14. Any current or chronic pain condition during the last year, located anywhere in the body
15. Allergy to capsaicin or hot peppers
16. Any skin lesion, breakage or irritation in the area targeted for the painful stimulus
17. Skin sensitivity to soaps/creams/perfumes or to heat
18. Poor circulation in the area targeted for the painful stimulus
19. Prior participation in a locomotor learning study in this lab within the last 2 years

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Digit Span Forward & Backward Test | the change between baseline and delivery (during application of intervention)
  number of digits (numbers) that can be repeated back in the same (DS forward) or the reverse (DS backward( order from which they were presented
Trail Making Test A & B | the change between baseline and delivery (during application of intervention)
  time required to draw a line connecting a series of numbers (TM-A) or a series of alternating letters and numbers (TM-B)

SECONDARY OUTCOMES:
Conner's Continuous Performance Test (CPT) 3 | the change between baseline and delivery (during application of intervention)
  response time for letters vs. 'x' stimuli; number of correct inhibited responses
Hopkins Verbal Learning Test- Revised | the change between baseline and delivery (during application of intervention)
  verbal memory for 3 semantic categories of 4 nouns each; immediate and delayed recall
Brief Visuospatial Memory Test- Revised | the change between baseline and delivery (during application of intervention)
  visual memory for 6 shapes and their location on a page; immediate and delayed recall and recognition
Stroop Test | the change between baseline and delivery (during application of intervention)
  response time and number of errors when stating the name of words printed in a congruent, neutral or incongruent color compared to the meaning of the words
Wisconsin Card Sorting Test | the change between baseline and delivery (during application of intervention)
  number of trials taken to deduce the new rule when the rules of a card game are changed without warning and without knowing what any of the rules are
Delis Kaplan Executive Functional System (D-KEFS) - Verbal Fluency Section | the change between baseline and delivery (during application of intervention)
  number of words stated that match a certain category or start with a certain letter in a given time period
NIH Toolbox Picture Sequence | the change between baseline and delivery (during application of intervention)
  reproduce the correct sequence of pictures
NIH Toolbox Flanker | the change between baseline and delivery (during application of intervention)
  response time and errors when asked to focus on a single visual stimulus amongst distractors
NIH Toolbox List Sorting | the change between baseline and delivery (during application of intervention)
  recall and sequencing of different visually and orally presented stimuli
NIH Toolbox Dimension Change Card Sort | the change between baseline and delivery (during application of intervention)
  errors selecting the correct dimension upon which to select a card, a cue for which is provided
NIH Toolbox Pattern Comparison | the change between baseline and during application of intervention
  errors and time required to determine whether several sets of two pictures are the same or not
Wechsler 4th ed - Spatial Addition | the change between baseline and delivery (during application of intervention)
  errors and time required to add or subtract the location of circles on a screen based on a given set of rules

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Morton, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States